CLINICAL TRIAL: NCT01369719
Title: Efficacy and Safety of Desferal Versus Osveral in Transfusional Iron Overload Patients With β-Thalassemia and Intermediate Thalassemia in Bandarabbas
Brief Title: Efficacy and Safety of Desferal Versus Osveral in Transfusional Iron Overload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Fariba Mansoori, Hormozgan University of Medical Sciences (HUMS)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Desferal versus Osveral
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2010-01

CONDITIONS: Thalassemia; Iron Overload; Transfusion Related Complications
Keywords: Thalassemia; Iron overload; transfusion; osveral; desferal
MeSH Terms: conditions — Thalassemia; Iron Overload | interventions — Deferasirox; Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osveral (Experimental): 20 mg/kg oral osveral daily
  Interventions: Drug: osveral
- desferal (Active Comparator): 40mg/kg desferal for 6 nights in a week subcutaneously
  Interventions: Drug: Desferal

INTERVENTIONS:
Drug: osveral — receive 20 mg/kg daily orally
  Other Names: deferasirox
  Arms: Osveral
Drug: Desferal — 40-50mg/Kg for 6 nights in each week subcutaneously
  Other Names: Deferoxamine
  Arms: desferal

SUMMARY:
Thalassemic patients often suffer from iron overload due to frequent blood transfusion. Oral iron chelators reduce iron overload in transfusion dependent patients. The aim of this study is to compare the efficacy and safety of osveral and desferal in transfusional iron overload patients with β-Thalassemia and intermediate Thalassemia in Bandarabbas.

DETAILED DESCRIPTION:
This is a double blinded randomized controlled trial on Efficacy and safety of Osveral and Desferal in thalassemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed intermedia or major thalassemia
* More then 2 years old
* Serum Ferritin level > 1000
* Normal Creatinine and Complete Blood Count (CBC)

Exclusion Criteria:

* HCV, HBV or HIV positive patients

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Ferritin level | 8 months
  ferritin level in months 4 and 8 of the study

SECONDARY OUTCOMES:
Hemoglobin level | 8 month
  hemoglobin level at months 4 and 8 off the study.
Drug side effects | 8 months
  Leuckopenia, thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Mansoori, Resident, Principal Investigator — Hormozgan University of Medical Sciences (HUMS)
Locations (1):
- Hormozgan University of Medical Sciences (HUMS), Bandar Abbas, Hormozgan, Iran